CLINICAL TRIAL: NCT01144494
Title: Circadian Rhythms of Aqueous Humor Dynamics in Subjects With Ocular Hypertension Using Brimonidine
Brief Title: Aqueous Humor Dynamics and Brimonidine
Acronym: Brimonidine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0220-10-FB; NCT01342419 (obsolete NCT alias)
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Intraocular Pressure
Keywords: Aqueous Humor Dynamics; Aqueous Humor Dynamics and Circadian Rhythms
MeSH Terms: interventions — Brimonidine Tartrate; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraocular pressure lowering drug (Active Comparator): Eyedrops for lowering intraocular pressure
  Interventions: Drug: Brimonidine
- Artificial Tears (Placebo Comparator): Lubricated eye drops
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Brimonidine — One drop of brimonidine in each eye three times a day for six weeks.
  Other Names: Mirvaso, Alphagan P
  Arms: Intraocular pressure lowering drug
Drug: Artificial tears — Lubricating drops added three times a day for six weeks
  Other Names: Systane
  Arms: Artificial Tears

SUMMARY:
This single-center, investigator-masked, crossover study is designed to investigate the circadian rhythms of aqueous humor dynamics in human subjects with ocular hypertension (OHT) before and after intervention with a commonly used ocular hypotensive medication, brimonidine for six weeks.

DETAILED DESCRIPTION:
Currently, the only effective treatment to prevent disease progression is lowering of the intraocular pressure (IOP).2 Usually, clinical IOP measurements are performed during the day with little information collected on nocturnal IOP. A recent surge of interest in nocturnal IOPs stems from the hypothesis that significant glaucomatous damage may occur at night.4,5 In response, some investigators have advocated particular classes of glaucoma medications based on their nocturnal IOP effects.6-8 The most efficacious drug on the market may not be the preferred treatment if it is ineffective at night. Therefore, the understanding of nighttime IOP and the aqueous humor dynamics that control it has important scientific, clinical, and commercial implications.

Previous research on glaucoma medications has been limited to the effects of ocular hypotensive drugs on 24-hour IOP or daytime aqueous humor dynamics. Few studies have evaluated nocturnal aqueous humor dynamics. The investigators recently completed studies of day and night differences in aqueous humor dynamics in patients treated with drugs from three different classes that include a prostaglandin analog, a beta blocker and a carbonic anhydrase inhibitor. The current study is designed to elucidate the physiological mechanisms driving the efficacy of brimonidine, an alpha 2 adrenergic agonist, throughout the 24-hour period, i.e. circadian rhythms in aqueous humor dynamics. Based on what the investigators know of 24 hour IOPs this drug is expected to work well at night potentially by enhancing uveoscleral outflow. This study will test this hypothesis.

This single-center, investigator-masked, crossover study is designed to investigate the circadian rhythms of aqueous humor dynamics in human subjects with ocular hypertension (OHT) before and after intervention with a commonly used ocular hypotensive medication, brimonidine. Thirty participants with ocular hypertension (intraocular pressure greater than 20mmHg) will be enrolled.

The subjects will undergo a baseline phase and medication phase using brimonidine. At both phases, they will attend a daytime and a nighttime study visit in which fluorophotometry will be used to calculate aqueous flow (production), trabecular outflow facility, and uveoscleral outflow. At the completion of the study, subjects will return to their previous ophthalmic clinic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 19 years of age or older
* Subjects must exhibit a history of untreated IOPs between 21 and 35 mmHg (inclusive)

Exclusion Criteria:

* Age less than nineteen years old
* Women who are pregnant, lactating or of childbearing potential who are not using birth control measures.
* Aphakia or pseudophakia
* Best corrected visual acuity worse than 20/60 in either eye
* Chronic or recurrent severe ocular inflammatory disease
* Ocular infection or inflammation within (3) months of screening visit.
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment.
* Any abnormality preventing reliable tonometry of either eye.
* Previous exposure to: beta-adrenergic antagonists, topical prostaglandin analogues within six (6) weeks of the baseline visit; α-adrenergic agonists within two (2) weeks of the baseline visit; and cholinergic agonists and carbonic anhydrase inhibitors within five (5) days of the treatment initiation visit.
* History of any severe ocular pathology (including severe dry eye) that would prelude the administration of a topical beta blocker, carbonic anhydrase inhibitor, or a topical prostaglandin.
* Any eye with a cup-to-disc ratio greater than 0.8.
* History of intraocular surgery
* History of ocular laser surgery
* History of severe or serious hypersensitivity to brimonidine or its vehicle.
* History of severe, unstable, or uncontrolled cardiovascular, hepatic or renal disease.
* History of bronchial asthma or chronic obstructive pulmonary disease (COPD).
* Less than one month (prior to baseline) stable dosing regimen of any non-glaucoma medication that would affect IOP.
* Gonioscopy angle < 2.
* Inability to be dosed with treatment medication
* Inability to discontinue contact lens wear.
* Therapy with any investigational agent within 30 days of screening.
* Use of any additional topical or systemic adjunctive ocular hypotensive medications during the study.
* History of open angle glaucoma (either primary open angle glaucoma or other cause of open angle glaucoma) or narrow angle glaucoma.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol B Toris, PhD, Principal Investigator — Research Instructor
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Fan S, Agrawal A, Gulati V, Neely DG, Toris CB. Daytime and nighttime effects of brimonidine on IOP and aqueous humor dynamics in participants with ocular hypertension. J Glaucoma. 2014 Jun-Jul;23(5):276-81. doi: 10.1097/IJG.0000000000000051. PMID 24886701

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects consented and then dropped out prior to assignment.
Groups:
- IOP Lowering Drug Then Art Tears: Eyedrops for lowering intraocular pressure
  Brimonidine: One drop of brimonidine in each eye three times a day for six weeks.
  Lubricated eye drops
  Artificial tears: Lubricating drops added three times a day for six weeks
- Artificial Tears Then IOP Lowering Drug: Lubricated eye drops
  Artificial tears: Lubricating drops added three times a day for six weeks
  Eyedrops for lowering intraocular pressure
  Brimonidine: One drop of brimonidine in each eye three times a day for six weeks.
Period: Overall Study
Arm/Group | IOP Lowering Drug Then Art Tears | Artificial Tears Then IOP Lowering Drug
Started | 15 | 18
Completed | 15 | 14
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: Intraocular pressure, episcleral venous pressure, and aqueous flow were calculated using data from 29 participants. However, tonography/outflow facility data on 2 participants were not reliable, therefore uveosleral outflow and outflow facility analysis were performed on 27 participants.
Groups:
- All Study Participants: participants were randomized to receive both IOP lowering drug and lubricating drops in a randomized order
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21
  African American | 6
  Hispanic | 1
  Native American | 1
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Seated Day-time IOP 9 am and 11 am, Supine Day-time IOP 9 am and 11 am, and Seated Night-time IOP 9 pm and 11 pm
Description: Seated day-time and supine day-time IOP was measured by pneumatonometer at 9 am and 11 am. Seated night-time IOP was measured at 9 pm and 11 pm.
Time Frame: 6 weeks
Population: some patients were consented but did not participate due to various reasons
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intraocular Pressure Lowering Drug | Artificial Tears
Number analyzed (Participants) | 29 | 29
mmHg
  Seated day-time 9 am | 18.1 (0.7) | 20.3 (0.7)
  Seated day-time 11 am | 18.0 (0.7) | 19.9 (0.8)
  Supine day-time 9 am | 23.1 (0.7) | 25.4 (0.7)
  Supine day-time 11 am | 23.1 (0.7) | 24.7 (0.8)
  Seated night-time 9 pm | 16.0 (0.6) | 18.0 (0.7)
  Seated night-time 11 pm | 16.7 (0.7) | 18.4 (0.7)

2. Primary Outcome: Supine Night-time & Day-time Seated Episcleral Venous Pressure (EVP)
Description: The episcleral venous pressure was measured using the episcleral venomanometer
Time Frame: 6 weeks plus 2 days
Population: some patients were consented but did not participate due to various reasons
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intraocular Pressure Lowering Drug | Artificial Tears
Number analyzed (Participants) | 27 | 27
mmHg
  Daytime Seated | 10.3 (0.2) | 10.3 (0.2)
  Nighttime Supine | 11.3 (0.3) | 11.2 (0.2)

3. Secondary Outcome: Aqueous Flow
Description: Measured by fluorophotometry during the day and night on 29 participants.
Time Frame: 6 weeks
Population: Measurements were taken in the day and night for each group and analysis was done comparing the difference between and within both groups in the day and night respectively.
  some patients were consented but did not participate due to various reasons
Measure: Mean (Standard Error); unit: µl/min
Groups:
- IOP Lowering Drug: Eyedrops for lowering intraocular pressure
  Brimonidine: One drop of brimonidine in each eye three times a day for six weeks.
Arm/Group | IOP Lowering Drug | Artificial Tears
Number analyzed (Participants) | 29 | 29
µl/min
  day-time measurement | 2.4 (0.1) | 2.3 (0.1)
  night-time measurement | 1.5 (0.1) | 1.5 (0.1)

4. Secondary Outcome: Uveoscleral Outflow
Description: Calculated from the modified Goldmann equation using data obtained at 9 am and 11 am. Goldmann equation involves data from aqueous flow, tonography/outflow facility, episcleral venous pressure and IOP. Tonography/outflow facility data on 2 participants were not reliable, therefore uveosleral outflow analysis was performed on 27 participants.
Time Frame: 6 weeks
Population: Tonography/outflow facility data on 2 participants were not reliable, therefore uveosleral outflow analysis was performed on 27 participants.
  some patients were consented but did not participate due to various reasons
Measure: Mean (95% Confidence Interval); unit: μL/min
Arm/Group | IOP Lowering Drug | Artificial Tears
Number analyzed (Participants) | 27 | 27
μL/min | 0.84 [0.24 to 1.46] | 0.72 [0.11 to 1.34]

5. Secondary Outcome: Outflow Facility
Description: Calculated from the measurement taken during the day and night. Tonography/outflow facility data was not reliable in 2 of the participants, therefore analysis was conducted on data from 27 participants.
Time Frame: 6 weeks
Population: Tonography/outflow facility data was not reliable in 2 of the participants, therefore analysis was conducted on data from 27 participants.
  some patients were consented but did not participate due to various reasons
Measure: Mean (Standard Error); unit: μL/min
Groups:
- IOP Lowering Drug (Day); IOP Lowering Drug (Night): Eyedrops for lowering intraocular pressure
  Brimonidine: One drop of brimonidine in each eye three times a day for six weeks.
- Artificial Tears (Day); Artificial Tears (Night): Lubricated eye drops
  Artificial tears: Lubricating drops added three times a day for six weeks
Arm/Group | IOP Lowering Drug (Day) | IOP Lowering Drug (Night) | Artificial Tears (Day) | Artificial Tears (Night)
Number analyzed (Participants) | 27 | 27 | 27 | 27
μL/min | 0.28 (0.02) | 0.28 (0.02) | 0.29 (0.02) | 0.29 (0.02)

ADVERSE EVENTS:
Arm/Group | Intraocular Pressure Lowering Drug | Artificial Tears
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 4/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraocular Pressure Lowering Drug (N=33) | Artificial Tears (N=33)
IOP equal to 35mmHg (Eye disorders) | 0 | 1
Acute anterior uveitis (Eye disorders) | 0 | 3
Corneal Epitheliopathy (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes